CLINICAL TRIAL: NCT06425549
Title: A Multicenter, Randomized, Parallel-Group, Double-Blind, Active-Controlled Study to Evaluate the Efficacy and Safety of Bimekizumab Compared to Ustekinumab in Children and Adolescents From 6 Years to Less Than 18 Years of Age With Moderate to Severe Plaque Psoriasis
Brief Title: A Study to Evaluate the Efficacy and Safety of Bimekizumab Compared to Ustekinumab in Children and Adolescents From 6 Years to Less Than 18 Years of Age With Moderate to Severe Plaque Psoriasis
Acronym: BE TOGETHER
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PS0021; U1111-1293-2383 (Other: WHO universal trial number (UTN)); 2023-503859-10-00 (Registry Identifier: CTIS (EU CT))
Record Dates: First submitted 2024-05-02; First posted 2024-05-22 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Moderate to Severe Plaque Psoriasis
Keywords: bimekizumab; BKZ; ustekinumab; paediatric study participants; children; adolescents; Psoriasis; PSO; Plaque Psoriasis; Paediatric Psoriasis; Pediatric Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — bimekizumab; Ustekinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- bimekizumab (Experimental): Study participants randomized to this arm receive bimekizumab dosage regimen 1 at pre-specified timepoints during the Initial Treatment Period (16 weeks). They continue to receive bimekizumab dosage regimen 2 in the Maintenance Period (32 weeks). Under certain conditions study participants may be offered to continue on bimekizumab dosage regimen 2 in the Open-label Extension (OLE) Period (104 weeks).
  Interventions: Drug: bimekizumab; Drug: placebo
- ustekinumab (Active Comparator): Study participants randomized to this arm receive ustekinumab at pre-specified timepoints during the Initial Treatment Period (16 weeks) and during the Maintenance Period. Under certain conditions participants may switch to bimekizumab dosage regimen 1 (16 weeks) and continue with bimekizumab dosage regimen 2 in the last 16 weeks of the Maintenance Period. Under certain conditions study participants may be offered to participate in the OLE Period also receiving bimekizumab dosage regimen 2.
  Interventions: Drug: bimekizumab; Drug: ustekinumab; Drug: placebo

INTERVENTIONS:
Drug: bimekizumab — Study participants receive bimekizumab (BKZ) administered as subcutaneous injection at pre-specified timepoints and dosage regimen during the study.
  Other Names: BKZ; UCB4940
Drug: ustekinumab — Study participants receive ustekinumab (USTE) administered as subcutaneous injection at pre-specified timepoints during the study.
  Other Names: USTE
  Arms: ustekinumab
Drug: placebo — Study participants receive placebo at pre-specified timepoints during the study to maintain the blinding.

SUMMARY:
The primary purpose of this study is to evaluate the efficacy of bimekizumab administered subcutaneously (sc) compared to active control (ustekinumab) in children and adolescents aged 6 to <18 years of age with moderate to severe plaque psoriasis (PSO).

ELIGIBILITY:
Inclusion Criteria:

* Study participant must be 6 to <18 years of age, inclusive, at the time of signing the informed consent/assent according to local regulation
* Study participant has had a diagnosis of moderate to severe plaque psoriasis (PSO) for at least 3 months prior to the Screening Visit
* Study participant meets the following at both the Screening and Baseline Visits:

  1. Body surface area (BSA) affected by PSO ≥10%
  2. . Investigator's Global Assessment (IGA) score ≥3 (on a scale from 0 to 4)
  3. . Psoriasis Area and Severity Index (PASI) score ≥12 OR

PASI score ≥10 plus at least 1 of the following:

i) Clinically relevant facial involvement ii) Clinically relevant genital involvement iii) Clinically relevant hand and foot involvement

* Study participant is a candidate for systemic PSO therapy and/or photo/chemotherapy and for treatment with ustekinumab per labeling
* Study participant has body weight ≥15 kg and body mass index for age percentile of ≥5 at Screening

Exclusion Criteria:

* Primary failure (no response within 12 weeks) to 1 or more interleukin-17 (IL-17) biologic response modifiers (eg, brodalumab, ixekizumab, secukinumab) OR more than 1 biologic response modifier other than an IL-17
* Study participant has a presence of guttate, inverse, pustular, or erythrodermic PSO or other dermatological condition that may impact the clinical assessment of PSO
* Study participant has a history of inflammatory bowel disease (IBD) or symptoms suggestive of IBD
* History of active tuberculosis unless successfully treated, latent TB unless prophylactically treated
* Study participant has an active infection or history of infections (such as serious infection, chronic infections, opportunistic infections, unusually severe infections)
* Study participant has previously received bimekizumab
* Study participant has previously received ustekinumab
* Study participant has received drugs outside the specified timeframes relative to the Baseline Visit or receives prohibited concomitant treatments
* Study participant has the presence of active suicidal ideation, or positive suicide behavior
* Study participant diagnosed with severe depression in the past 6 months (prior to Screening) should be excluded
* Study participant has a history of psychiatric inpatient hospitalization within the past year before enrolling into the study

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 168 (Estimated)
Dates: Start 2024-06-25 (Actual); Primary Completion 2028-08-21 (Estimated); Study Completion 2030-11-08 (Estimated)

PRIMARY OUTCOMES:
Psoriasis Area Severity Index 90 (PASI90) response at Week 16 | Week 16
  The PASI90 response assessments are based on at least 90% improvement in the PASI score from Baseline. This is a scoring system that averages the redness, thickness, and scaliness of the psoriatic lesions (on a 0-4 scale), and weights the resulting score by the area of skin involved. Body divided into 4 areas: head, arms, trunk to groin, and legs to top of buttocks. Assignment of an average score for the redness, thickness, and scaling for each of the 4 body areas with a score of 0 (clear) to 4 (very marked). Determining the percentage of skin covered with PSO for each of the body areas and converting to a 0 to 6 scale. Final PASI= average redness, thickness, and scaliness of the psoriatic skin lesions, multiplied by the involved psoriasis area score of the respective section, and weighted by the percentage of the person's affected skin for the respective section. The minimum possible PASI score is 0= no disease, the maximum score is 72= maximal disease.
Investigator´s Global Assessment (IGA) 0/1 response at Week 16 | Week 16
  The Investigator's Global Assessment (IGA) measures the overall psoriasis severity following a 5-point scale (0-4), where scale 0= clear, no signs of psoriasis; presence of post-inflammatory hyperpigmentation, scale 1= almost clear, no thickening; normal to pink coloration; no to minimal focal scaling, scale 2= mild, just detectable to mild thickening; pink to light red coloration; predominately fine scaling, 3= moderate, clearly distinguishable to moderate thickening; dull to bright red; moderate scaling and 4= severe, severe thickening with hard edges; bright to deep dark red coloration; severe/coarse scaling covering almost all or all lesions.
  IGA response (Clear or Almost Clear) is defined as clear [0] or almost clear [1] with at least a two-category improvement from Baseline.

SECONDARY OUTCOMES:
PASI75 response at Week 4 | Week 4
  The PASI75 response assessments are based on at least 75% improvement in the PASI score from Baseline. This is a scoring system that averages the redness, thickness, and scaliness of the psoriatic lesions (on a 0-4 scale), and weights the resulting score by the area of skin involved. Body divided into 4 areas: head, arms, trunk to groin, and legs to top of buttocks. Assignment of an average score for the redness, thickness, and scaling for each of the 4 body areas with a score of 0 (clear) to 4 (very marked). Determining the percentage of skin covered with PSO for each of the body areas and converting to a 0 to 6 scale. Final PASI= average redness, thickness, and scaliness of the psoriatic skin lesions, multiplied by the involved psoriasis area score of the respective section, and weighted by the percentage of the person's affected skin for the respective section. The minimum possible PASI score is 0= no disease, the maximum score is 72= maximal disease.
PASI100 response at Week 16 | Week 16
  A PASI100 responder is defined as a subject that achieves 100% reduction from Baseline in the PASI score. This is a scoring system that averages the redness, thickness, and scaliness of the psoriatic lesions (on a 0-4 scale), and weights the resulting score by the area of skin involved. Body divided into 4 areas: head, arms, trunk to groin, and legs to top of buttocks. Assignment of an average score for the redness, thickness, and scaling for each of the 4 body areas with a score of 0 (clear) to 4 (very marked). Determining the percentage of skin covered with PSO for each of the body areas and converting to a 0 to 6 scale. Final PASI= average redness, thickness, and scaliness of the psoriatic skin lesions, multiplied by the involved psoriasis area score of the respective section, and weighted by the percentage of the person's affected skin for the respective section. The minimum possible PASI score is 0= no disease, the maximum score is 72= maximal disease.
PASI90 response at Week 48 | Week 48
  The PASI90 response assessments are based on at least 90% improvement in the PASI score from Baseline. This is a scoring system that averages the redness, thickness, and scaliness of the psoriatic lesions (on a 0-4 scale), and weights the resulting score by the area of skin involved. Body divided into 4 areas: head, arms, trunk to groin, and legs to top of buttocks. Assignment of an average score for the redness, thickness, and scaling for each of the 4 body areas with a score of 0 (clear) to 4 (very marked). Determining the percentage of skin covered with PSO for each of the body areas and converting to a 0 to 6 scale. Final PASI= average redness, thickness, and scaliness of the psoriatic skin lesions, multiplied by the involved psoriasis area score of the respective section, and weighted by the percentage of the person's affected skin for the respective section. The minimum possible PASI score is 0= no disease, the maximum score is 72= maximal disease.
IGA 0/1 response at Week 48 | Week 48
  The Investigator's Global Assessment (IGA) measures the overall psoriasis severity following a 5-point scale (0-4), where scale 0= clear, no signs of psoriasis; presence of post-inflammatory hyperpigmentation, scale 1= almost clear, no thickening; normal to pink coloration; no to minimal focal scaling, scale 2= mild, just detectable to mild thickening; pink to light red coloration; predominately fine scaling, 3= moderate, clearly distinguishable to moderate thickening; dull to bright red; moderate scaling and 4= severe, severe thickening with hard edges; bright to deep dark red coloration; severe/coarse scaling covering almost all or all lesions.
  IGA response (Clear or Almost Clear) is defined as clear [0] or almost clear [1] with at least a two-category improvement from Baseline.
PASI100 response at Week 48 | Week 48
  A PASI100 responder is defined as a subject that achieves 100% reduction from Baseline in the PASI score. This is a scoring system that averages the redness, thickness, and scaliness of the psoriatic lesions (on a 0-4 scale), and weights the resulting score by the area of skin involved. Body divided into 4 areas: head, arms, trunk to groin, and legs to top of buttocks. Assignment of an average score for the redness, thickness, and scaling for each of the 4 body areas with a score of 0 (clear) to 4 (very marked). Determining the percentage of skin covered with PSO for each of the body areas and converting to a 0 to 6 scale. Final PASI= average redness, thickness, and scaliness of the psoriatic skin lesions, multiplied by the involved psoriasis area score of the respective section, and weighted by the percentage of the person's affected skin for the respective section. The minimum possible PASI score is 0= no disease, the maximum score is 72= maximal disease.
IGA 0 response at Week 16 | Week 16
  The Investigator's Global Assessment (IGA) measures the overall psoriasis severity following a 5-point scale (0-4), where scale 0= clear, no signs of psoriasis; post-inflammatory hyperpigmentation may be present, scale 1= almost clear, no thickening; normal to pink coloration; no to minimal focal scaling, scale 2= mild, just detectable to mild thickening; pink to light red coloration; predominately fine scaling, 3= moderate, clearly distinguishable to moderate thickening; dull to bright red; moderate scaling and 4= severe, severe thickening with hard edges; bright to deep dark red coloration; severe/coarse scaling covering almost all or all lesions.
  IGA 0 response (Clear) is defined as clear [0] with at least a two-category improvement from Baseline.
IGA 0 response at Week 48 | Week 48
  The Investigator's Global Assessment (IGA) measures the overall psoriasis severity following a 5-point scale (0-4), where scale 0= clear, no signs of psoriasis; post-inflammatory hyperpigmentation may be present, scale 1= almost clear, no thickening; normal to pink coloration; no to minimal focal scaling, scale 2= mild, just detectable to mild thickening; pink to light red coloration; predominately fine scaling, 3= moderate, clearly distinguishable to moderate thickening; dull to bright red; moderate scaling and 4= severe, severe thickening with hard edges; bright to deep dark red coloration; severe/coarse scaling covering almost all or all lesions.
  IGA 0 response (Clear) is defined as clear [0] with at least a two-category improvement from Baseline.
Incidence of treatment-emergent adverse events (TEAE)s | From Baseline (Week 0) to End of Safety Follow-up (up to Week 164)
  An adverse event (AE) is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product, which does not necessarily have a causal relationship with this treatment. Treatment-emergent AEs are defined as those AEs that have a start date on or following the first dose of IMP through the final dose of IMP + 20 weeks.
Incidence of serious TEAEs | From Baseline (Week 0) to End of Safety Follow-up (up to Week 164)
  An serious adverse event (SAE) must meet 1 or more of the following criteria:
  * Results in death
  * Is life-threatening
  * Requires inpatient hospitalization or prolongation of existing hospitalization
  * Results in persistent disability/incapacity
  * Is a congenital anomaly/birth defect
  * Important medical event that, based upon appropriate medical judgment, may jeopardize the patient or subject and may require medical or surgical intervention to prevent 1 of the other outcomes listed in the definition of serious.
  Treatment-emergent AEs are defined as those AEs that have a start date on or following the first dose of IMP through the final dose of IMP + 20 weeks.
Incidence of TEAEs leading to discontinuation of Investigational Medicinal Product (IMP) | From Baseline (Week 0) to End of Safety Follow-up (up to Week 164)
  An adverse event (AE) is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product, which does not necessarily have a causal relationship with this treatment. Treatment-emergent AEs are defined as those AEs that have a start date on or following the first dose of IMP through the final dose of IMP + 20 weeks. This measure considers any TEAE leading to permanent discontinuation of IMP regardless of reason.
Incidence of TEAEs leading to withdrawal from the study | From Baseline (Week 0) to End of Safety Follow-up (up to Week 164)
  An adverse event (AE) is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product, which does not necessarily have a causal relationship with this treatment. Treatment-emergent AEs are defined as those AEs that have a start date on or following the first dose of IMP through the final dose of IMP + 20 weeks. This measure considers any TEAE leading to permanent withdrawal from study.
Incidence of TEAEs predefined as safety topics of interest | From Baseline (Week 0) to Week 48 and to End of Safety Follow-up (up to Week 164)
  Safety topics of interest are infections (serious, opportunistic, fungal, and tuberculosis), inflammatory bowel disease, and injection site reactions.
Change from Baseline in vital signs (systolic blood pressure) | From Baseline (Week 0) up to Week 48
  Blood pressure will be measured in millimeters of mercury (mmHg).
Change from Baseline in vital signs (diastolic blood pressure) | From Baseline (Week 0) up to Week 48
  Blood pressure will be measured in millimeters of mercury (mmHg).
Change from Baseline in vital signs (pulse rate) | From Baseline (Week 0) up to Week 48
  Pulse rate will be measured in beats per minute (beats/min).
Incidence of clinically significant physical examination findings reported as TEAEs | From Baseline (Week 0) up to Week 48
  Clinically significant findings or worsening of previous findings since the physical examination at Baseline will be reported as TEAEs.
Change from Baseline in height (growth assessment) | From Baseline (Week 0) up to Week 48
  Growth assessment, as assessed by the change from Baseline in height.
Change from Baseline in weight (growth assessment) | From Baseline (Week 0) up to Week 48.
  Growth assessment, as assessed by the change from Baseline in weight.
Change from Baseline in hematology parameters (platelet count) | From Baseline (Week 0) up to Week 48
  Platelets will be measured in number of platelets per liter (10^9/L).
Change from Baseline in hematology parameters (erythrocytes) | From Baseline (Week 0) up to Week 48
  Erythrocytes will be measured in number of red blood cells per liter (10^12/L).
Change from Baseline in hematology parameters (hemoglobin) | From Baseline (Week 0) up to Week 48
  Hemoglobin will be measured in grams per liter (g/L).
Change from Baseline in hematology parameters (hematocrit) | From Baseline (Week 0) up to Week 48
  Hematocrit will be measured in volume percentage (%) of red blood cells in blood.
Change from Baseline in biochemistry parameters (alkaline phosphatase, alanine aminotransferase, aspartate aminotransferase, gamma-glutamyltransferase) | From Baseline (Week 0) up to Week 48
  Alkaline phosphatase, alanine aminotransferase, aspartate aminotransferase and gamma-glutamyltransferase will be measured in units per liter (U/L).
Change from Baseline in hematology parameters (basophils, eosinophils, lymphocytes, monocytes, neutrophils, leukocytes) | From Baseline (Week 0) up to Week 48
  Basophils, eosinophils, lymphocytes, monocytes, neutrophils and leukocytes will be measured in number of white blood cells per liter (10^9/L).
Change from Baseline in biochemistry parameters (glucose, potassium, sodium, calcium) | From Baseline (Week 0) up to Week 48
  Glucose, potassium, sodium and calcium will be measured in millimoles per liter (mmol/L).
Change from Baseline in biochemistry parameters (total bilirubin and direct bilirubin, total protein, blood urea nitrogen, and creatinine) | From Baseline (Week 0) up to Week 48
  Clinical chemistry parameters will be measured in micromols per liter (μmol/L).
Change from Baseline in Children's Dermatology Life Quality Index (CDLQI) total score at Week 16 | Week 16, compared to Baseline
  The CDLQI is a questionnaire designed to measure the impact of skin diseases on the lives of children. The questionnaire consists of 10 questions that are based on the experiences of children with skin disease. The instrument asks participants about symptoms and feelings, leisure, school or holidays, personal relationships, sleep, and treatment. The questions relate to the impact of the skin disease on the child over the last week. The CDLQI total score ranges from 0 to 30 with higher scores indicating higher impact of skin disease on quality of life (Qol).
Change from Baseline in Children's Dermatology Life Quality Index (CDLQI) total score at Week 48 | Week 48, compared to Baseline
  The CDLQI is a questionnaire designed to measure the impact of skin diseases on the lives of children. The questionnaire consists of 10 questions that are based on the experiences of children with skin disease. The instrument asks participants about symptoms and feelings, leisure, school or holidays, personal relationships, sleep, and treatment. The questions relate to the impact of the skin disease on the child over the last week. The CDLQI total score ranges from 0 to 30 with higher scores indicating higher impact of skin disease on quality of life (Qol).
Change from Baseline in Childhood Health Assessment Questionnaire (CHAQ) disability index at Week 16 for study participants with juvenile PsA prior to Baseline | Week 16, compared to Baseline
  The CHAQ is a questionnaire designed to capture physical function in children and adolescents with juvenile rheumatoid arthritis. The CHAQ comprises 2 indices, Disability and Discomfort. The Disability Index assesses the degree of difficulty experienced over the past week across 30 items in the following 8 categories of the daily living activities: dressing and grooming, arising, eating, walking, hygiene, reach, grip, and activities. The Disability Index ranges from 0 (no disability) to 3 (maximum disability). Discomfort is determined by the presence of pain, as measured by a 100-mm visual analogue scale (VAS). In addition, a final global assessment item asks study participants to rate how they are doing by placing a mark on a 100 mm VAS.
Change from Baseline in Peak Pruritus numerical rating scale (NRS) score at Week 16 | Week 16, compared to Baseline
  The Peak Pruritus NRS measures the worst level of itching in the past 24 hours on an 11-point scale ranging from 0 (no itch) to 10 (worst imaginable itch).
Plasma bimekizumab concentrations prior to and following IMP administration over the Initial Treatment Period, over the Maintenance Period, and over the OLE Period | From Baseline to End of OLE Period (up to 144 weeks)
  Plasma bimekizumab concentrations prior to investigational medicinal product (IMP) administration and following investigational medicinal product (IMP) administration
Plasma anti-bimekizumab antibodies prior to and following IMP administration over the Initial Treatment Period, over the Maintenance Period, and over the OLE Period | From Baseline to End of OLE Period (up to 144 weeks)
  Anti-bimekizumab antibody (AbAb) detection prior to investigational medicinal product (IMP) administration and following investigational medicinal product (IMP) administration

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273
Locations (50):
- United States (9):
  - Ps0021 50162, Fountain Valley, California
  - Ps0021 50161, Los Angeles, California
  - Ps0021 50196, Northridge, California
  - Ps0021 50581, Miami, Florida
  - Ps0021 50344, Indianapolis, Indiana
  - Ps0021 50599, Kew Gardens, New York
  - Ps0021 50084, Charleston, South Carolina
  - Ps0021 50201, Arlington, Texas
  - Ps0021 50355, Dallas, Texas
- Belgium (2):
  - Ps0021 40121, Brussels
  - Ps0021 40420, Liège
- Canada (3):
  - Ps0021 50618, Mississauga
  - Ps0021 50357, St. John's
  - Ps0021 50617, St. John's
- Ps0021 40748, Plzen-bory, Czechia
- France (2):
  - Ps0021 40742, Argenteuil
  - Ps0021 40754, Nantes
- Germany (10):
  - Ps0021 40740, Bad Bentheim
  - Ps0021 40515, Berlin
  - Ps0021 40138, Bonn
  - Ps0021 40356, Dresden
  - Ps0021 40023, Erlangen
  - Ps0021 40645, Frankfurt am Main
  - Ps0021 40758, Hamburg
  - Ps0021 40249, Kiel
  - Ps0021 40747, Mainz
  - Ps0021 40177, Münster
- Hungary (3):
  - Ps0021 40746, Debrecen
  - Ps0021 40744, Kaposvár
  - Ps0021 40745, Szeged
- Italy (4):
  - Ps0021 40440, Ancona, Località Torrette
  - Ps0021 40749, Catania
  - Ps0021 40085, Pisa
  - Ps0021 40567, Roma
- Japan (3):
  - Ps0021 20071, Nagasaki
  - Ps0021 20033, Nagoya
  - Ps0021 20337, Shimotsuga-gun
- Poland (8):
  - Ps0021 40741, Bialystok
  - Ps0021 40625, Lodz
  - Ps0021 40832, Lodz
  - Ps0021 40091, Nowa Sól
  - Ps0021 40737, Rzeszów
  - Ps0021 40743, Szczecin
  - Ps0021 40334, Wroclaw
  - Ps0021 40738, Wroclaw
- Spain (5):
  - Ps0021 40750, Alicante
  - Ps0021 40159, Barcelona
  - Ps0021 40751, Esplugues de Llobregat
  - Ps0021 40752, Granada
  - Ps0021 40753, Santiago de Compostela

IPD SHARING:
Plan to Share IPD: Yes
Data from this study may be requested by qualified researchers six months after product approval in the US and/or Europe, or global development is discontinued, and 18 months after trial completion. Investigators may request access to anonymized IPD and redacted study documents which may include: raw datasets, analysis-ready datasets, study protocol, blank case report form, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a pre-specified time, typically 12 months, on a password protected portal. This plan may change if a determination is made that the data cannot be adequately anonymized.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data from this study may be requested by qualified researchers six months after product approval in the US and/or Europe or global development is discontinued, and 18 months after trial completion.
Access Criteria: Qualified researchers may request access to anonymized IPD and redacted study documents which may include: raw datasets, analysis-ready datasets, study protocol, blank case report form, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a pre-specified time, typically 12 months, on a password protected portal.
URL: https://Vivli.org